CLINICAL TRIAL: NCT05366868
Title: Durable Effect of Imeglimin on the Glycemic Control in Patients With Type 2 Diabetes Mellitus: a Multicenter, Open-label, Randomized, Controlled Trial (DIGNITY Trial)
Brief Title: Durable Effect of Imeglimin on the Glycemic Control in Patients With Type 2 Diabetes Mellitus
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: National Center for Global Health and Medicine, Japan (Other Government)
Collaborators: Sumitomo Pharma Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Kohjiro Ueki, Director, Diabetes Research Center, Research Institute, National Center for Global Health and Medicine, Japan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 004371; jRCTs051180211 (Registry Identifier: jRCT)
Record Dates: First submitted 2022-04-15; First posted 2022-05-09 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — imeglimin; Metformin; Vildagliptin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Imeglimin (Experimental): Imeglimin 1000 mg orally twice daily in the morning and evening (2000 mg daily).
  Interventions: Drug: Imeglimin
- Metformin (Active Comparator): Metformin 500 mg orally twice daily in the morning and evening (1000 mg daily). However, until 2 weeks after the start of treatment, 250 mg should be administered orally twice daily in the morning and evening. Thereafter, after 4, 8, or 12 weeks, the dose may be increased up to 750 mg twice daily (1500 mg daily) if the physician determines that the hypoglycemic effect is inadequate.
  Interventions: Drug: Metformin
- Vildagliptin (Active Comparator): Vildagliptin 50 mg orally twice daily in the morning and evening (100 mg daily).
  Interventions: Drug: Vildagliptin

INTERVENTIONS:
Drug: Imeglimin — Imeglimin 1000 mg orally twice daily in the morning and evening (2000 mg daily).
  Arms: Imeglimin
Drug: Metformin — Metformin 500 mg orally twice daily in the morning and evening (1000 mg daily). However, until 2 weeks after the start of treatment, 250 mg should be administered orally twice daily in the morning and evening. Thereafter, after 4, 8, or 12 weeks, the dose may be increased up to 750 mg twice daily (1500 mg daily) if the physician determines that the hypoglycemic effect is inadequate.
  Arms: Metformin
Drug: Vildagliptin — Vildagliptin 50 mg orally twice daily in the morning and evening (100 mg daily).
  Arms: Vildagliptin

SUMMARY:
Study subjects will be randomly assigned to the three groups and receive the study drug for maximum of 156 weeks and undergo blood samplings and other diabetes mellitus-related tests. The aim of the present study is to evaluate the durability of glycemic control over 3 years for patients with type 2 diabetes on diet and exercise therapy treated with oral hypoglycemic drug monotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with type 2 diabetes mellitus who are 20 years of age or older at the time of obtaining consent.
2. Patients being treated with diet and exercise therapy only at the time of eligibility test However, if the patient is taking one oral hypoglycemic drug at the time of obtaining consent, the patient must be able to wash out the oral hypoglycemic drug for at least 12 weeks before the start of study treatment.
3. Patients whose HbA1c level is between 7.0% and 9.0% as measured at the time of the eligibility test.
4. Patients who have given written consent to participate in this study.

Exclusion Criteria:

When consent is obtained

1. Patients with type 1 diabetes mellitus
2. Patients who have been given more than 2 oral hypoglycemic drugs within 12 weeks
3. Patients who have received glucagon like peptide-1 receptor agonist (short-term use of insulin for trauma or educational admission) within 1 year or less
4. Patients with proliferative retinopathy (except for patients with stable treated proliferative retinopathy)
5. Patients with severe diabetic neuropathy (patients with severe symptoms and significant support for daily life)
6. Patients with a contraindication to Imeglimin, Metformin, or Vildagliptin
7. Patients with severe obesity (BMI 35 kg/m^2 or more)
8. Patients with NYHA (New York Heart Association) cardiac function classification of Grade III or IV within 1 year of evaluation
9. Excessive regular drinkers
10. Patients with a previous history of lactic acidosis
11. Patients with severe cachexia, diabetic coma or precoma
12. Patients with severe infections, surgical patients and those with serious injuries
13. Patients who are pregnant, who are planning to be pregnant, or who are breastfeeding
14. Patients who are undergoing treatment for malignancy or those with a history of treatment for malignancy within 5 years
15. Patients who are participating in a clinical study with other interventions
16. Patients to whom a responsible physician/investigator judged inappropriate for participating in the study In case of eligibility testing
17. Patients with an estimated glomerular filtration rate(eGFR) of 45 mL/min/1.73m^2 or less including those undergoing dialysis
18. Patients with severe hepatic disorders (Child-Pugh classification Grade C)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 567 (Estimated)
Dates: Start 2022-05-26 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Time from study drug initiation (Week 0) to detection of two consecutive HbA1c levels of 7.0% or higher by laboratory tests after Week 16. | From 16 to 156 weeks after the start of study drug administration

SECONDARY OUTCOMES:
Time from Week 0 to addition of a type 2 diabetes mellitus medication after Week 16 | From 16 to 156 weeks after the start of study drug administration
Time from detection of two consecutive HbA1c levels of 7.0% or higher to addition of a type 2 diabetes mellitus medication after Week 16. | From 16 to 156 weeks after the start of study drug administration
HbA1c level, fasting blood glucose level, and their changes from baseline at each measurement point | From 0 to 156 weeks after the start of study drug administration
Maximum decrease in HbA1c level during the observation period | From 0 to 156 weeks after the start of study drug administration
Proportion of patients achieving HbA1c level less than 7.0% at each measurement point | From 0 to 156 weeks after the start of study drug administration
Number of times of achieving HbA1c level less than 7.0% during the observation period | From 0 to 156 weeks after the start of study drug administration
Time from Week 0 to detection of two consecutive HbA1c levels of 7.0% or higher by laboratory tests after Week 16 by patient characteristics | From 0 to 156 weeks after the start of study drug administration

CONTACTS AND LOCATIONS:
Overall Officials: Kohjiro Ueki, M.D., Ph.D., Principal Investigator — Center Hospital of the National Center for Global Health and Medicine
Locations (1):
- Center Hospital of the National Center for Global Health and Medicine, Shinjuku-Ku, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: Undecided